CLINICAL TRIAL: NCT02206386
Title: Homecare Agency-Randomized Trial of Web Implementation Strategy for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH096441 (NIH); R01MH096441 (NIH)
Record Dates: First submitted 2014-07-25; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MentalHealthTraining-Net (Experimental): MHTraining-Net is an implementation strategy that uses a web-based platform with several long distance tools (e.g. e-learning modules, consultation, telephone calls, toolkits, and discussion boards) to deliver four types of implementation activities: infrastructure development, training and education, quality improvement, and social networking.
  Interventions: Other: MHTraining-Net
- Enhanced Support (Active Comparator): Nurses in agencies randomized to Enhanced Support have full access to the study protocol and to recorded trainings in the use of the protocol and depression screening posted by Brightree.
  Interventions: Other: Enhanced Support

INTERVENTIONS:
Other: MHTraining-Net — See Arm Description for more details.
  Arms: MentalHealthTraining-Net
Other: Enhanced Support — Nurses in agencies randomized to Enhanced Support have full access to the study protocol and to recorded training in the use of the protocol and depression screening posted by Brightree.
  Arms: Enhanced Support

SUMMARY:
To identify effective implementation strategies that can efficiently promote the use of evidence-based practices (EBP) across a large number of geographically dispersed, independent Home Health Agencies (HHAs). This study will use an agency-randomized design to test the effectiveness of a web-based implementation strategy (MHTraining-Net) on the use of an evidence-based practice for geriatric depression by home healthcare agencies. The EBP is known as the Depression CARE for PATients at Home (CAREPATH) Intervention. The effectiveness of MHTraining-Net will be measured by an agency's adherence to the Depression CAREPATH protocol with its depressed patients and changes in their patients' depressive symptoms over the episode of care.

DETAILED DESCRIPTION:
MHTraining-Net uses a web-based platform and several long distance tools (e.g., e-learning modules, telephone or web consultation, telephone calls, toolkits, and discussion boards) to deliver four types of implementation activities: infrastructure development, training and education, quality improvement, and social networking. MHTraining-Net was developed to ensure that the Depression CAREPATH (CARE for PATients at Home), specifically, and evidence-based practices, generally, can be implemented widely and successfully across independent organizations within a sector of care.

PROCEDURES: The effectiveness of MHTraining-Net on the implementation of the Depression CAREPATH will be tested in an agency-randomized trial of 160 HHAs. All HHAs are clients of Brightree (formerly CareAnyware, Inc), a software company that offers web-based point-of-care clinical management and administrative support for HHA nationwide. HHA clinicians record relevant data that is transmitted directly to Brightree for clinical and administrative purposes, including quality improvement initiatives. As part of each HHA's contract with Brightree is permission for using these data for performance enhancement research.

Brightree has already programmed Cornell's Depression CAREPATH, a depression care management protocol, into its clinical management system so that all nurses use the protocol. To promote the use of the protocol, Brightree has posted two relevant videos (archived Patient Health Questionnaire-9 training web seminar training); demonstration of how to navigate the protocol within the software) on its user education website.

Brightree will randomize HHAs to either MHTraining-Net, (N=100) or to Enhanced Support (N=60). Enhanced Support will have access to only the two training videos until the end of the study when they will be invited to MHTraining-Net. These procedures represent Brightree's typical "roll-out" approach on introducing new training and products to their client HHAs.

The study will test its hypotheses using three sets of data:

1. Summary statistics describing the size and type of the 160 HHAs as well as their average nurse productivity over the 12 months preceding and following the study;
2. Routinely collected administrative data on patients age >65 who screen positive for depression over one year, including Medicare-mandated assessments, medication lists, transaction files, indicators of whether the depression care management protocol was used, and Medicare case-mix adjustment and reimbursement indicators. We are using to term 'patients' to refer to a full episode of patient care, defined from the Start-of-Care date to Discharge, recognizing that a small proportion of unique individuals may have more than one full episode of care. We will not be able to identify such individuals. These data will be aggregated at the patient level in preparation for performance enhancement analyses using Brightree's routine procedures. Brightree will code the data, remove identifiers, and transmit them to Weill Cornell on a regular basis using the Weill Cornell ITS Department secure servers and protocols.
3. Agency-level data on the use of the MHTraining-Net website (e.g., summary reports on 'hits' of each webpage) and agency-initiated contacts (telephone, email) through records maintained by Cornell project staff.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients 65 and older
* Patients screened for depression using the Patient Health Questionnaire-2

Exclusion Criteria:

* Geriatric patients under age 65
* Patients who were not screened for depression using the Patient Health Questionnaire-2

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7800 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Nurse adherence to the depression care management protocol (Depression CAREPATH intervention). | one episode (60 days)
  At least one follow-up depression assessment and evidence of case coordination (e.g., contacting the patient's physician or a specialist) to evaluate treatment needs.

SECONDARY OUTCOMES:
Patient reduction in depression symptoms | one episode of care (60 days)
  Patient Health Questionnaire (two item version and nine item version)

CONTACTS AND LOCATIONS:
Overall Officials: Martha L Bruce, PhD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, White Plains, New York, United States

REFERENCES:
- [Background] Bruce ML, Raue PJ, Sheeran T, Reilly C, Pomerantz JC, Meyers BS, Weinberger MI, Zukowski D. Depression Care for Patients at Home (Depression CAREPATH): home care depression care management protocol, part 2. Home Healthc Nurse. 2011 Sep;29(8):480-9. doi: 10.1097/NHH.0b013e318229d75b. PMID 21881429
- [Background] Bruce ML, Sheeran T, Raue PJ, Reilly CF, Greenberg RL, Pomerantz JC, Meyers BS, Weinberger MI, Johnston CL. Depression care for patients at home (Depression CAREPATH): intervention development and implementation, part 1. Home Healthc Nurse. 2011 Jul-Aug;29(7):416-26. doi: 10.1097/NHH.0b013e31821fe9f7. PMID 21716043